CLINICAL TRIAL: NCT05539040
Title: Understanding the Role of Right Atrial Ectopy-triggering Ganglionated Plexuses in Atrial Fibrillation
Brief Title: The Role of Right Atrial Ectopy Triggering Ganglionated Plexuses in AF
Acronym: RGanglia-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA2481; 314366 (Other: IRAS)
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Arrhythmia; Atrial Fibrillation
Keywords: Atrial Fibrillation; Ganglionated plexus; Arrhythmia; Cardiology; Right atrium; Ectopy; Electrophysiology; GP; AF
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Intervention Model Description: This will be a single centre pilot study with a control arm and outcomes will be measured prospectively on both an intention-to-treat and per-protocol basis.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Right atrial GP ablation in addition to pulmonary vein isolation
  Interventions: Procedure: Right Atrial ganglionated plexus ablation; Diagnostic Test: Holter Monitor; Procedure: Pulmonary vein isolation; Diagnostic Test: Personal ECG recordings; Other: Quality of life questionnaire
- Control (Active Comparator): PVI alone with no GP mapping or ablation
  Interventions: Diagnostic Test: Holter Monitor; Procedure: Pulmonary vein isolation; Procedure: Right cavo-tricuspid and left roof linear ablation; Diagnostic Test: Personal ECG recordings; Other: Quality of life questionnaire

INTERVENTIONS:
Procedure: Right Atrial ganglionated plexus ablation — A 3D electroanatomic map of the right atrium will be made. During sinus rhythm, the ablation catheter will be positioned at a spot to test with HFS. The right atrium will be paced at a fixed rate, for up to four beats to ensure that there is no ventricular capture then a short burst of HFS will be synchronized to each paced stimulus for up to 15 trains. This will be performed using a custom-built GP stimulator that has been validated for reproducibility against Grass Stimulator (AstroMed).
  All Sites will be marked on the 3D map and the positive sites will be ablated at the end of the mapping. If the patient converts to AF, then DC cardioversion will be performed. If mapping in sinus rhythm is not feasible, HFS will be performed continuously for several seconds to identify atrioventricular dissociating GPs (AVD-GPs).
  Every ablated GP site will be re-tested with HFS at the end of the procedure until they are all rendered non-functional.
  Arms: Intervention
Diagnostic Test: Holter Monitor — 48 hour Holter monitors will be performed post procedure to monitor for recurrence of AF.
  These will be performed at 3, 6, 9, 12 months
Procedure: Pulmonary vein isolation — Transseptal puncture for access into the left atrium will be guided by TOE and fluoroscopy.
  ACT will be maintained at 300s with heparin. A 3D electroanatomic map of the left atrium will be created and all PVs will be identified. Touch-up radiofrequency ablation will be performed at electrical gaps around the reconnected PVs until complete PVI is achieved.
Procedure: Right cavo-tricuspid and left roof linear ablation — CONTROL ARM (Redo-PVI) only: If all Pulmonary veins are isolated at the start of the procedure, the operator will be allowed to perform a right cavo-tricuspid and left roof linear ablation.
  Arms: Control
Diagnostic Test: Personal ECG recordings — All patients will be provided with an AliveCor KardiaMobile-6L ECG recorder. The device will continue to be used within its CE-marked and NICE-approved purpose. Patients will be asked to take a daily recording from this, once the blanking period is over, in addition to taking a recording if symptomatic. Patients will submit this to the connected care team at Hammersmith Hospital via a secure NHS.net email address, who will assess the recordings both for the study and clinical purposes.
Other: Quality of life questionnaire — A Quality of life questionnaire will be performed at baseline, 6 and 12 months to assess the effect of the procedures on patients quality of life.

SUMMARY:
Atrial fibrillation (AF) is the most common rhythm disturbance of the heart. It can affect people of any age but usually happens as we get older. It can cause palpitations, breathlessness, lethargy, and fainting attacks. It is also associated with an increased risk of strokes.

The best treatment for it at the moment involves burning or freezing (ablation) the heart muscle in a part of the heart called the left atrium. The ablation injures the heart muscle around the so-called pulmonary veins and the procedure is called a 'pulmonary vein isolation'. This procedure work in about 60% of people.

The study team have found that there are nerve endings in the heart that also cause AF and have shown that ablating these nerve endings also prevents AF. These Nerve endings are known as ganglionated plexuses (GPs).

The study team would now like to perform a trial in people who still have AF after the usual pulmonary vein procedure. The study team hope that ablating the nerve endings that cause AF (GPs), we will stop their AF coming back. The study team will compare this procedure to the normal approach of doing the pulmonary vein isolation again

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disturbance and causes physical discomfort and strokes.

The the best long-term treatment of AF is catheter ablation in a part of the heart called the left atrium and works in about 60-70% of patients.

The study team have discovered that that there are nerve endings in the heart that cause AF (GP sites). The study team have previously treated patients with AF by ablating these nerve endings (GP ablation) in a part of the heart called the left atrium.

The study team have treated patients with AF by ablation of these nerve ending in the left atrium. The treatment worked in a similar number of people to the standard treatment but caused less heart injury than the standard treatment

There are similar nerve endings in another part of the heart called the right atrium. The study team want to find out if ablating these nerve endings in the right atrium can help people for whom the standard treatment in the left atrium has not worked.

STUDY PROTOCOL: The study will run at at one hospital (Hammersmith Hospital). The study team will look at the information on patients who have been placed on the waiting list for an AF ablation. The study team will approach patients who have previously had an ablation and coming back for another procedure.

Patients will be given information about the study and discuss the issues with the research team. Patients who decide to participate will be allocated an anonymised number and their information included on a research database and will be encrypted for use only by the research team.

Patients in the study will be randomly assigned to one of two treatment pathways. All patients will then continue with their standard NHS treatment to prepare them for the procedure. All patients will have all the steps of the ablation done in the same way, including the repeat pulmonary vein isolation procedure which they have been advised to have by their own doctor.

The group of patients allocated to receive right sided ablation to treat the nerve endings procedure will have this done in addition to the repeat pulmonary vein isolation.

The study team will aim to recruit 116 patients to the study. All patients will stop any heart rhythm medication prior to the procedure. A 48 hour heart rhythm monitor will be obtained prior to patients' procedure. The study team will also ask patients to complete a survey to assess their quality of life.

All patients will have their procedures under general anaesthesia. An ultrasound from inside the oesophagus will be used to exclude blood clot in the heart. Access to the heart will be through the veins in the leg and transeptal puncture to get into the left atrium. All patients will first undergo a repeat pulmonary vein isolation. 3D mapping software will be used to identify the pulmonary veins and then these will be isolated from the rest of the heart by using radiofrequency energy to burn the tissue which connects these areas to the rest of the heart. This will be the end of the procedure for those patients receiving standard treatment.

The patients allocated to right atrial GP ablation will then have map of the right atrium created and the sites which contains the nerves supplying the heart identified. These will be found using high-frequency electrical stimulation delivered by a custom-built stimulator that has been shown to be comparable to the existing technology. When the sites of these nerves are found, they will be marked on the map of the right atrium and then they will undergo ablation with radiofrequency energy till they are no longer detectable.

If the patient is not in a normal rhythm before or during the procedure, then they may require an electric shock to return them to normal. The procedures in each arm will take between 2hrs and 3hrs to perform

Follow Up:

All heart rhythm medication patient used to take before ablation will be continued during the 3 months after procedure, except for amiodarone. After 3 months, patients will stop all heart rhythm medication if they are well and free of symptoms or AF.

At 3, 6, 9, 12 months following patients' procedures, 48hour heart monitors will be fitted or implanted devices will be reviewed, to assess if any atrial fibrillation has happened. The Quality of life survey will be repeated at 6 and 12 months after the ablation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females from 18 to 85yrs old
* Symptomatic paroxysmal atrial fibrillation
* Suitable candidate for catheter ablation
* Signed informed consent

Exclusion Criteria:

* Contraindication to catheter ablation
* Contraindication for general anaesthetic
* Presence of a left ventricular thrombus
* Valvular disease that is grade moderate or greater
* Any form of cardiomyopathy
* Severe cerebrovascular disease
* Active gastrointestinal bleeding
* Serum Creatinine >200umol/L/ on dialysis/ at risk of dialysis
* Active infection or fever
* Life expectancy shorter than the duration of the trial
* Allergy to contrast
* Moderate to severe heart failure and/or NYHA Class III-IV
* Bleeding or clotting disorders or inability to receive heparin
* Uncontrolled diabetes (HbA1c ≥73mmol/mol or HbA1c ≤64mmol/mol and Fasting Blood Glucose ≥9.2mmol/L)
* Malignancy needing therapy
* Pregnancy or women of childbearing potential not using a highly effective method of contraception
* Unable to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
atrial arrhythmia lasting >30secs | 1 year
  Any recorded atrial arrhythmia lasting >30seconds will meet the primary endpoint for the trial.

SECONDARY OUTCOMES:
Complications | 1 year
  Number of patients experiencing a procedural complication.
Usage of antiarrhythmic drugs | 1 year
  number of patients using antiarrhythmic drugs to control symptoms and pathology of AF
Quality of life questionnaire | 1 year
  Quality of life will be assess pre and post procedure to assess if any improvement has been seen post procedure. An increase in the AFEQT questionnaire score will reflect a decrease in quality of life
Re-do procedures | 1 year
  number of repeat procedures will be assessed and compared between the to arms
Radiofrequency time | day of the procedure.
  The quantity of radiofrequency ablation in each arm of the trail will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, MBBChir, PhD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data with other researchers